CLINICAL TRIAL: NCT05037552
Title: Additional Benefit of Hemostatic Sealant in Preservation of Ovarian Reserve During Laparoscopic Ovarian Cystectomy
Brief Title: Benefit of Hemostatic Sealant in Preservation of Ovarian Reserve
Acronym: FLOKIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RECHMPL20_0664
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Benign Ovarian Cyst; Cystectomy
Keywords: Ovarien cyst; Bipolar; Ovarian reserve; Hemostatic agent; Coelioscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BIPOLAR FORCEPS (Active Comparator): The bipolar forceps allow electrocoagulation and are part of the standard laparoscopy box, delivered by the sterilization service to the gynecology operating room.
  Interventions: Procedure: Bipolar coagulation
- FLOSEAL (Experimental): FLOSEAL® is a hemostatic agent based on gelatin of bovine origin added to thrombin of human origin. It is a recommended medical device in surgical procedures as an adjunct to hemostasis when control of bleeding, arterial jet seepage, ligation or any other conventional method proves impractical or ineffective.
  During this study, it will be used in 1st intention.
  Interventions: Procedure: Coagulation by FLOSEAL haemostatic agent

INTERVENTIONS:
Procedure: Bipolar coagulation — Cystectomy will be done via laparoendoscopic surgery After identifying the correct plane of cleavage, the stripping technique will be used. The cyst wall will be gently pulled down from the remaining ovary with two pairs of atraumatic forceps.
  Once the whole cyst wall will be separated from the ovary cortex, bleeding of the remaining ovarian stromal tissue will be controlled by bipolar coagulation. Then, the remnant tissue will be examined using irrigation and coagulated with minimal bipolar power (20-W current) on any sites that are bleeding.
  Arms: BIPOLAR FORCEPS
Procedure: Coagulation by FLOSEAL haemostatic agent — Cystectomy will be done via laparoendoscopic surgery After identifying the correct plane of cleavage, the stripping technique will be used. The cyst wall will be gently pulled down from the remaining ovary with two pairs of atraumatic forceps.
  Once the whole cyst wall will be separated from the ovary cortex, bleeding of the remaining ovarian stromal tissue will be controlled by either hemostatic sealants (FloSeal). Using a laparoscopic applicator, FloSeal will be applied to the surface of bleeding sites under direct vision and the ovarian cortex was gently pressed for 2 min with small gauze.
  Arms: FLOSEAL

SUMMARY:
Introduction : The most common technique used for ovarian cystectomy is the stripping technique. After stripping the cyst wall, the subsequent bleeding of the ovarian stromal wound is usually controlled by bipolar coagulation or/and by suturing. However, hemostasis achieved with bipolar coagulation could result in damage to the ovarian reserve. To avoid damage to healthy ovarian tissue, hemostasis using various topical hemostatic agents has been introduced to control post- cystectomy ovarian wound bleeding. Among these, FloSeal (Baxter Healthcare Corporation, Deer- field, IL, USA) is a hemostatic sealant composed of a gelatin-based matrix and thrombin solution.

Aim: The aim of the study is to evaluate the impact of topical hemostatic sealants and bipolar coagulation during laparoscopic ovarian benign cyst resection on ovarian reserve by comparing the rates of decrease in anti- Müllerian hormone (AMH).

Methods: A randomized prospective data collection was made on women aged 18-45 years who planned to have laparoscopic ovarian cystectomy at one of two institutions (n = 80), Montpellier University Hospital and Nimes University Hospital, France. Patients were randomly divided into two groups treated with either a topical hemostatic sealant (Floseal) or bipolar coagulation for hemostasis. Preoperative, 3-month and 6-month postoperative AMH levels were checked and the rates of decrease of AMH were compared.

ELIGIBILITY:
Inclusion Criteria:

* Cyst diameter between 3 and 10cm
* Preoperative AMH level >0,5ng/ml
* Understanding and acceptance of the protocol

Exclusion Criteria:

* Post-menopausal status
* Any suspicious finding of malignant ovarian disease
* Change of contraception method leading to AMH variation
* Allergy to bovine products found before inclusion
* Pregnancy
* Patient who has already participated in the protocol
* Person deprived of liberty by judicial or administrative decision
* Person protected by law, under tutorship or curatorship
* Patient participating in another interventional research on the human person in progress
* Refusal of participation after a period of reflection
* Patient not affiliated or beneficiary of a national health insurance system

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Serum anti-Mullerian hormone (AMH) level preoperative | Between 2 and 17 days before cystectomy
  A biological assessment with determination of the serum AMH level will be carried out for each patient during the preoperative consultation.
Serum anti-Mullerian hormone (AMH) level at 3 months | 3 months after the cystectomy
  A biological assessment with determination of the serum AMH level will be carried out for each patient, 3 months postoperatively.
Serum anti-Mullerian hormone (AMH) level at 6 months | 6 months after the cystectomy
  A biological assessment with determination of the serum AMH level will be carried out for each patient, 6 months postoperatively.

SECONDARY OUTCOMES:
Time to achieve hemostasis | From the end of the cystectomy to the end of hemostasis (up to 1 hour)
  The time is measured in minutes from the end of the cystectomy to the end of hemostasis.
Use of additional hemostatsis technique | From the end of the cystectomy to the end of hemostasis, during surgery
  Another technique can be used to achieve hemostasis: bipolar forceps, suture or second hemostasis agent. The other technique will be specified if it is used
Blood loss | From the start of the surgery to the end of hemostasis
  Blood loss will be measured in ml throughout the surgery.
Intraoperative adverse effects | From the end of the cystectomy to the end of hemostasis
  Adverse effects related to the coagulation procedure will be collected.
Revision surgery for bleeding at the operative site | From the end of the cystectomy to the end of hemostasis
  In the event of bleeding at the operative site, revision surgery may be necessary. In this case the information will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Martha DURAES, MD, Study Director — Montpellier University Hospital
Locations (2):
- France (2):
  - CHU de Montpellier, Montpellier
  - CHU de Nîmes, Nîmes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FLOSEAL user guide — http://www.baxter.ca/sites/g/files/ebysai1431/files/2018-11/Floseal_EN_FR.pdf